CLINICAL TRIAL: NCT04274478
Title: Biofeedback to Reduce Freezing of Gait in Parkinson Patients - Ceriter/Insole Parkinson Disease (IPD)-1
Brief Title: Adaptive Auditive Cueing As a Therapy for Freezing of Gait in Parkinson Patients
Acronym: BioFOGP-IPD1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Non CE-certified status of device
Sponsor: Ceriter Nederland BV (Industry)
Collaborators: Ziekenhuis Oost Limburg (ZOL) Hospital Genk, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BioFOGP-IPD-1-ZOL
Record Dates: First submitted 2020-02-02; First posted 2020-02-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single group (Other)
  Interventions: Device: Auditive cueing

INTERVENTIONS:
Device: Auditive cueing — Based on gait measurement, auditive cueing is generated automatically to check its impact on patients with Freezing Of Gait.

SUMMARY:
The first goal of the study is to investigate whether an algorithm can reliably detect Freezing of Gait (FOG) in Parkinson patients based on participant gait data generated by a pressure insole. The second goal is to investigate whether Auditive Cueing (AC) based on such a detection reduces the frequency and length of FOG episodes in those participants.

The study will be conducted per Good Clinical Practice principles.

ELIGIBILITY:
Inclusion Criteria:

* must have more than 1 FOG episode/day
* must be patient in Ziekenhuis Oost Limburg (ZOL)

Exclusion Criteria:

* not able to speak Dutch
* cannot give informed consent (mental health)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-04-11 (Actual)

PRIMARY OUTCOMES:
The F1-score of FOG detection from the measured and classified (normal walk vs FOG) gait data compared to manually scored recorded video. | 8 walks are performed in 1 hospital visit within 4 weeks of enrollment. Total assessment time estimate is 2x 30 minutes.
  The participants perform 4 walks without AC on standardized tracks while being video-recorded. During the walks, gait data is recorded and then scored (for each time point) by the algorithm into normal walk or FOG. The video recording is scored manually according to the criteria as described in reference Gilat. M. and represents the true state of walking.
  The F1-score is calculated from the algorithm scoring vs the manual scoring: a True Positive is true freezing which is classified by the algorithm as freezing. A True Negative is a true normal walk which is classified as a normal walk. Similarly, a False Positive is a true normal walk which is classified as FOG and a False Negative is a true FOG which is classified as a normal walk.
  The same 4 walks are performed both in OFF and in ON. OFF measurement is only performed when the PI has given permission to do so. ON measurement is performed 1 hour after taking their standard medication.
The change in the number of FOG-episodes with and without AC | 1 week after the first hospital visit (for Outcome 1).
  The participants again perform 4 walks in OFF and in ON but now with AC.
  The average number of freezing episodes is calculated for each participant in OFF and in ON with and without AC. The change between the average without AC and the average with AC is calculated as well as its level of significance. These changes are computed for each walk, for each individual participant across all walks and across all participants.
The change in the total duration of FOG-episodes with and without AC | within 1 to 3 weeks after the first hospital visit
  The participants again perform 4 walks in OFF and in ON but now with AC.
  The average duration of freezing episodes is calculated in the same way as their number per Outcome 2.

SECONDARY OUTCOMES:
The sensitivity of FOG detection from the measured and classified (normal walk vs FOG) gait data compared to manually scored recorded video. | Within 4 weeks of enrollment
  Same data collection as for outcome 1. Sensitivity is calculated from the algorithm scoring vs the manual scoring.
The specificity of FOG detection from the measured and classified (normal walk vs FOG) gait data compared to manually scored recorded video. | within 1 to 3 weeks after the first hospital visit
  Same data collection as for outcome 1. Specificity is calculated from the algorithm scoring vs the manual scoring.

CONTACTS AND LOCATIONS:
Overall Officials: An Driesen, MD, Neurologist, Principal Investigator — ZOL Genk
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naghavi N, Miller A, Wade E. Towards Real-Time Prediction of Freezing of Gait in Patients With Parkinson's Disease: Addressing the Class Imbalance Problem. Sensors (Basel). 2019 Sep 10;19(18):3898. doi: 10.3390/s19183898. PMID 31509999
- [Background] Nonnekes J, Janssen AM, Mensink SH, Oude Nijhuis LB, Bloem BR, Snijders AH. Short rapid steps to provoke freezing of gait in Parkinson's disease. J Neurol. 2014 Sep;261(9):1763-7. doi: 10.1007/s00415-014-7422-8. Epub 2014 Jun 24. PMID 24957299
- [Background] Barthel C, Nonnekes J, van Helvert M, Haan R, Janssen A, Delval A, Weerdesteyn V, Debu B, van Wezel R, Bloem BR, Ferraye MU. The laser shoes: A new ambulatory device to alleviate freezing of gait in Parkinson disease. Neurology. 2018 Jan 9;90(2):e164-e171. doi: 10.1212/WNL.0000000000004795. Epub 2017 Dec 20. PMID 29263221
- [Background] Zach H, Janssen AM, Snijders AH, Delval A, Ferraye MU, Auff E, Weerdesteyn V, Bloem BR, Nonnekes J. Identifying freezing of gait in Parkinson's disease during freezing provoking tasks using waist-mounted accelerometry. Parkinsonism Relat Disord. 2015 Nov;21(11):1362-6. doi: 10.1016/j.parkreldis.2015.09.051. Epub 2015 Oct 1. PMID 26454703
- [Background] Ginis P, Heremans E, Ferrari A, Bekkers EMJ, Canning CG, Nieuwboer A. External input for gait in people with Parkinson's disease with and without freezing of gait: One size does not fit all. J Neurol. 2017 Jul;264(7):1488-1496. doi: 10.1007/s00415-017-8552-6. Epub 2017 Jun 26. PMID 28653213
- [Background] Gilat M. How to Annotate Freezing of Gait from Video: A Standardized Method Using Open-Source Software. J Parkinsons Dis. 2019;9(4):821-824. doi: 10.3233/JPD-191700. PMID 31524181